CLINICAL TRIAL: NCT05829616
Title: A Phase I, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Initial Antitumor Activity of QLS12004 in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of QLS12004 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS12004-101
Record Dates: First submitted 2023-03-23; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS12004 (Experimental): Subjects will be treated with different dose groups of QLS12004 according to the frequency and periodicity of administration as specified in the protocol, until disease progression or unacceptable toxicity.
  Interventions: Drug: QLS12004

INTERVENTIONS:
Drug: QLS12004 — Subjects will be treated with different dose groups of QLS12004 according to the frequency and periodicity of administration as specified in the protocol, until disease progression or unacceptable toxicity.

SUMMARY:
This study is a single-arm, open, dose-escalation, and dose-expansion phase I clinical trial of QLS12004 in patients with advanced solid tumors, designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of QLS12004 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a single-arm, open, dose-escalation, and dose-expansion phase I clinical trial of QLS12004 in patients with advanced solid tumors, designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of QLS12004 in subjects with advanced solid tumors.The frequency of administration and the dose to be administered in subsequent clinical studies will be determined based on a combination of preliminary data.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF);
2. Age ≥ 18 years when ICF is signed;
3. At least one target lesion as defined per RECIST Version (v) 1.1;
4. Dose escalation phase: Pts with histologically or cytologically confirmed advanced solid tumors, who have failed standard therapy or for whom no standard therapy is available;
5. Dose escalation phase: HR+/HER2-advanced breast cancer that has failed prior CDK4/6 inhibitor combined with endocrine therapy;
6. Eastern Cooperative Oncology Group performance status of 0 or 1;
7. Adequate hematologic and organ function;
8. Female subjects who are not pregnant or breastfeeding
9. Male and female subjects able to have children must agree to use highly effective method of contraception throughout the study and for at least 90 days after last dose.

Exclusion Criteria:

1. Subjects with major cardiovascular and cerebrovascular diseases;
2. Any condition that required systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication ≤ 14 days before the first dose of study drug;
3. Subjects who have received chemotherapy, endocrine therapy, immunotherapy, and targeted therapy, other anti-tumor treatments, or participating in other clinical studies is less than 4 weeks before the first administration of investigational product;
4. Known psychiatric or substance abuse disorders that would interfere with the requirements of the study;
5. HIV-positive or syphilis spiral antibody-positive persons;
6. Major organ surgery (excluding puncture biopsy) or significant trauma within 4 weeks prior to the first dose, or the need for elective surgery during the trial;
7. Known hypersensitivity to the test drug or any of its excipients;
8. History or current evidence of any condition, therapy, or laboratory abnormality, that might confound the results of the trial, or interfere with the participant's participation for the full duration of the study, or investigators/sponsor consider the subjects are not suitable for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-17 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
AEs, TEAEs, TRAEs, SAEs | up to 2 years
  Incidence, severity and relevance to the trial drug of adverse events (AEs), treatment-related adverse events (TEAEs), treatment-related adverse events (TRAEs) and serious adverse events (SAEs)
DLT | Up to 21 days after the first dose
  Dose-limiting toxicity
MTD | Up to 21 days after the first dose
  maximum tolerated dose
RP2D | Up to 21 days after the first dose
  recommended phase II dose

SECONDARY OUTCOMES:
Tmax | up to 2 years
  Time to Reach Maximum (peak) Plasma Concentration Following Drug Administration
Cmax | up to 2 years
  Maximum Plasma Drug Concentration
ORR | up to 2 years
  Objective Response Rate
DCR | up to 2 years
  Disease Control Rate
PFS | up to 2 years
  Progression-free Survival
OS | up to 2 years
  Objective Response Rate

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of the General Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No